CLINICAL TRIAL: NCT02127736
Title: Pharmacological Conditioning of Sleep Patterns in Healthy Participants Using Amitriptylin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winfried Rief (Other)
Responsible Party: Sponsor-Investigator, Winfried Rief, Prof. Dr. Winfried Rief, Philipps University Marburg
Organization: Philipps University Marburg (Other)
Other Study IDs: PSG40
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Amitriptyline

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Amitriptyline; Drug: Placebo
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline
  Arms: Experimental group
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate whether an Amitriptylin induced change in sleep patterns can be conditioned according to learning theory in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 years to 69 years
* willingness to refrain from alcohol consumption throughout the study
* regular sleeping habits
* fluent in German language
* is not dependent on driving to get to the study center
* provide written informed consent
* ability to understand the explanations and instructions given by the study physician and the investigator

Exclusion Criteria:

* Contraindications to study medication intake according to the information sheet for health professionals (Summary of medicinal Product Characteristics, SmPC) assessed by physical examination (including ECG) and medical history

  * allergies to amitriptyline hydrochloride or any of its ingredients
  * acute intoxication with alcohol, analgetics, hypnotics or any other psychotropic drug
  * urinary retention
  * delirium
  * untreated closed-angle glaucoma
  * prostatic hyperplasia
  * pyloric stenosis
  * paralytic ileus
  * suicidal thoughts
  * liver/ kidney/ pulmonary insufficiency
  * myasthenia gravis
  * hypokalemia
  * bradycardia
  * coronary heart disease, cardiac arrhythmias, long QT syndrome or other clinically relevant cardiac disorders
  * increased risk of seizures/ history of seizures
  * substance dependence syndrome/ history of substance dependence syndrome
* Allergies to ingredients of placebo or novel-tasting drink (CS)
* currently pregnant (verified by urine pregnancy test) or lactating
* patients suffering from a mental disorder as verified by the International Diagnosis Checklists (IDCL)
* patients suffering from a medical condition (assessed by the study physician)
* Concomitant medication interfering with study medication intake due to potential interactions
* participation in any other clinical trial 3 months prior to visit 1
* employee of the Sponsor or the principal investigator

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Objective Total Sleep Time | 5 nights during the study
  assessed by polysomnography
Percentage of rapid eye movement (REM) sleep | 5 nights during the study
  assessed by polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

REFERENCES:
- [Derived] Rheker J, Rief W, Doering BK, Winkler A. Assessment of adverse events in clinical drug trials: Identifying amitriptyline's placebo- and baseline-controlled side effects. Exp Clin Psychopharmacol. 2018 Jun;26(3):320-326. doi: 10.1037/pha0000194. PMID 29863388